CLINICAL TRIAL: NCT05993949
Title: Phase 1b Study of Brexucabtagene Autoleucel Plus Dasatinib in Adults With Acute Lymphoblastic Leukemia
Brief Title: Study of Brexucabtagene Autoleucel Plus Dasatinib in Adults With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-68603; NCI-2023-05591 (Registry Identifier: NCI- Clinical Trial Reporting Program)
Record Dates: First submitted 2023-07-10; First posted 2023-08-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lymphoblastic Leukemia
Keywords: Leukemia; CAR T cell therapy; Brexucabtagene Autoleucel; Dasatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib (Experimental): Oral dasatinib 100mg
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 3 pulses of oral dasatinib (100 mg daily) beginning on Day 4 (+up to 2 days) for 3 days (with 4 days off), repeated weekly. The weekly 3-day pulse schedule of dasatinib may continue for up to 3 months in subjects who continue to meet the dasatinib eligibility criteria and who do not meet off treatment/off study criteria

SUMMARY:
To assess the feasibility of oral dasatinib pulses (3 consecutive days per week) during the first month following infusion of brexucabtagene autoleucel (Tecartus) in adults with relapsed or refractory B-cell acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-precursor ALL defined as one of the following:

  * Primary refractory disease (>=5% blasts or persistent extramedullary disease following induction therapy)
  * First or later relapse of marrow or extramedullary disease
  * Persistence of MRD defined as detectable ALL by flow cytometry, PCR, or next-generation sequencing
  * Relapsed or refractory disease after allogeneic transplant provided individual is at least 100 days from transplant at time of enrollment
  * Patients with isolated, asymptomatic CNS relapse will be eligible

    * Age >=18 years
    * Eastern cooperative oncology group (ECOG) performance status of 0-2
    * Adequate renal, hepatic, pulmonary and cardiac function defined as:
  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 cc/min
  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dl, except in individuals with Gilbert's syndrome.
  * Cardiac ejection fraction ≥ 50%, no evidence of clinically significant pericardial effusion, and no clinically significant arrhythmias
  * Baseline oxygen saturation > 92% on room air
  * QTc ≤ 500ms

    * In individuals previously treated with blinatumomab, CD19 tumor expression in bone marrow or peripheral blood by flow cytometry or extramedullary site by IHC or flow cytometry
    * Negative serum or urine beta-HCG test in females of childbearing potential within 3 weeks of enrollment
    * Subjects of childbearing or child fathering potential must be willing to practice birth control from the time of enrollment on this study Page 10 of 83 Version 1.0 dated 27-April-2023 and for six (6) months after receiving the preparative conditioning regimen.
    * Must be able to give informed consent. Legal authorized representative (LAR) is permitted if subject is cognitively able to provide verbal assent.

Exclusion Criteria:

* History of dasatinib intolerance
* Known sensitivity or allergy to aminoglycosides or any agents/reagents used in this study
* Blast count > 75% in the bone marrow.
* History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 2 years
* Presence of CNS-3 disease with neurological changes
* History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage with clinical signs or symptoms
* History of concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond or any known bone marrow failure syndrome
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
* Primary immunodeficiency
* Known infection with HIV, hepatitis B (HBsAg positive) or untreated hepatitis C virus
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
* Salvage chemotherapy including TKIs for Ph+ ALL within 1 week prior to enrollment
* Pregnant or breast feeding
* Patients with known autoimmune disease requiring the use of systemic immunosuppressive therapy within the last year
* Corticosteroid therapy within 7 days prior to enrollment
* Acute or chronic GVHD requiring systemic treatment within 4 weeks prior to enrollment
* Live vaccine ≤ 4 weeks prior to enrollment
* Any medical condition that in the judgement of the investigator is likely to interfere with assessment of safety or efficacy of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of dasatinib pulses | 1 month
  Feasibility of administering oral dasatinib pulses (3 consecutive doses per week) during the first month following Tecartus infusion. Feasibility will be defined as the ability of 8 out of 20 subjects to miss no more than one cycle (defined as one week of at least three consecutive days of dasatinib) within the first month following Tecartus infusion.

SECONDARY OUTCOMES:
Safety of oral dasatinib pulses | 2 years
  Defined by a description of adverse events and serious adverse events at least possibly related to dasatinib following CAR T cell therapy; it will include an analysis of the sequential toxicity boundaries in that the analysis does not lead to a pause in the study; further defined as no reports of suspected death on study.
Overall response rate | 3 months
  The definitions for response are primarily based on the standardized response criteria defined by National Comprehensive Cancer Network (NCCN) Guidelines (NCCN, 2021 v.2).
Complete Response (CR) | 3 months
  The definitions for response are primarily based on the standardized response criteria defined by National Comprehensive Cancer Network (NCCN) Guidelines (NCCN, 2021 v.2).
MRD-negative Complete Response (CR) | 3 months
  The definitions for response are primarily based on the standardized response criteria defined by National Comprehensive Cancer Network (NCCN) Guidelines (NCCN, 2021 v.2).
Duration of CR in responders | 2 years
Progression Free Survival (PFS) following Tecartus plus dasatinib | 2 years
  PFS is defined as the time from the start of the investigational therapy to the date of radiographic progression
Overall Survival (OS) following Tecartus plus dasatinib | 2 years
  OS is defined as the time from the date of initial disease diagnosis to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Lori Muffly, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States